CLINICAL TRIAL: NCT03977610
Title: The Role of Ga68-PSMA-11 PET Imaging in Prostate Cancer Patients Undergoing Androgen Deprivation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jing-Ren Tseng, Nuclear Medicine, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201801384A0
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Prostate Cancer
Keywords: Prostate cancer; Androgen deprivation therapy; Ga-68 PSMA Ligand; Treatment response
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ga68-PSMA ligand (Experimental): Glass vial with 4~20 mCi(148-740 MBq) of 68Ga-PSMA ligand in ≤10% EtOH with aqueous sterile water for injection solution (approximately 15.5 mL), more than 0.33 mCi/mL @ EOS; One time dose of 2-5 mCi (74-185 MBq) for PET Imaging ; i.v. injection
  Interventions: Drug: Ga-68 PSMA ligand

INTERVENTIONS:
Drug: Ga-68 PSMA ligand — For PSMA PET/CT scan, the subject will have catheter(s) placed for intravenous administration of [68Ga]PSMA-11. Subjects will receive a single intravenous bolus of 2-5 mCi [68Ga]PSMA-11 and received PET/CT scan 60 minutes later. Patient will underwent two times of PSMA-11 PET/CT scans before and under androgen deprivation therapy within a 10-14 weeks interval.
  Other Names: Ga68-PSMA-11 (Gallium-68 labeled HBED-CC PSMA)

SUMMARY:
This is an open-label single arm clinical trial, Plan to enroll approximately a total of 43 evaluable subjects. According to the estimated missing rate 15%, the sample size in this study is 51.

Inclusion criteria:

To be eligible for inclusion, each patient must fulfill all of the following criteria:

1. Males with 40-85 years of age and life expectancy more than 3 months
2. Pathology-proved prostate cancer patients and classified as clinical stage III or IV (including lymph node or bone metastasis)
3. Willing to sign the informed consent

Exclusion criteria:

Patient who has any of the following criteria will be excluded from the trial:

1. Unable to tolerate the PET/CT scan, such as those with claustrophobia, unable to lie still, consciousness unclear, vital sign unstable.
2. With renal impairment (glomerular filtration rate lower than 30 ml/min/1.73 m2), and allergy to medium contrast.
3. Significant abnormal lab data (AST or ALT more than three times of normal value), and high risk to conduct examination after evaluations of PI.
4. Patient had previous malignancy history
5. Patient had known allergy history or is probably allergy to Ga68-PSMA-11

DETAILED DESCRIPTION:
It is a single-arm clinical trial. The primary endpoint is diagnostic positivity rate of Ga68-PSMA-11 in metastasis lesion. Sample size calculation is performed using two-sided one-proportion test to achieving an 82% power at the 5% level of significance. The primary measurement of positivity can be obtained for the one-proportion test with statistical hypotheses H0: P = P0 versus H1: P≠P0. We assume the alternative positivity rate is 65.9% and the null positivity rate is 43.9% which is the reference value from Maurer T et al (J Urol. 2016;195:1436-1443). Thus, the sample size needed is 43. According to the estimated missing rate 15%, the sample size in this study is 51. The sample size calculation was performed using PASS software (Power Analysis and Sample Size version 11.0.8, NCSS, Kaysville, Utah, USA). All subjects enrolled must meet eligibility criteria based on the inclusion/exclusion criteria detailed in Section 5.4 and 5.5.

For PET/CT PSMA scan, the subject will have catheter(s) placed for intravenous administration of [68Ga]PSMA-11. Subjects will receive a single intravenous bolus of 2-5 mCi [68Ga]PSMA-11 and received PET/CT scan 60 minutes later. The data acquisition begin with non-contrast CT at 120kVp, automated mAs, and a pitch of 1.5, followed by PET acquisition from the mid-thigh to skull-base, 3 minutes each bed. After image acquisition, the subject will be observed for half an hour, and will be discharged if no adverse event happens. EKG, blood and biochemistry test will be performed before and after scan no more than two weeks. Patient will underwent two times of PSMA-11 PET/CT scans before and under androgen deprivation therapy within a 10-14 weeks interval. In the follow up period, if metastatic castration-resistance status happens, patient may underwent optional PSMA-11 PET/CT scan by attending's discrimination in order to give appropriate treatment suggestions.

Time elapsed from the last PSA determination until PET scan was no more than 6 weeks in all patients. Patients will receive complementary workups. All of the images were interpreted by a team of two nuclear medicine physicians and one radiologist. In cases of questionable findings, the decision was made by consensus of at least two observers using pre-specified criteria. For patients with discrepancy image findings between each modality, biopsy results may be taken into consideration to determine the final status.

ELIGIBILITY:
Inclusion Criteria:

1. Males with 40-85 years of age and life expectancy more than 3 months
2. Pathology-proved prostate cancer patients and classified as clinical stage III or IV (including lymph node or bone metastasis)
3. Willing to sign the informed consent

Exclusion Criteria:

1. Unable to tolerate the PET/CT scan, such as those with claustrophobia, unable to lie still, consciousness unclear, vital sign unstable.
2. With renal impairment (glomerular filtration rate lower than 30 ml/min/1.73 m2), and allergy to medium contrast.
3. Significant abnormal lab data (AST or ALT more than three times of normal value), and high risk to conduct examination after evaluations of PI.
4. Patient had previous malignancy history
5. Patient had known allergy history or is probably allergy to Ga68-PSMA-11

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Change of lesion detection number by PET imaging | 10-14 weeks
  Lesion detection number before and under androgen deprivation therapy on the PSMA PET imaging with a time interval 10-14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Ren Tseng, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital ,Linkou, Taoyuan, Taiwan